CLINICAL TRIAL: NCT00205465
Title: A Randomized, Double-Blind, Placebo-Controlled, Safety and Tolerability Study of VX-765 in Subjects With Chronic Plaque Psoriasis Requiring Systemic Therapy
Brief Title: Phase 2 Clinical Study in Psoriasis With Oral Investigational Drug VX-765
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Robert Kauffman, M.D., Ph.D, Vertex Pharmaceuticals Incorporated
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VX04-765-301
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — belnacasan

INTERVENTIONS:
Drug: VX-765

SUMMARY:
To evaluate the safety and tolerability of VX-765 in subjects with chronic plaque psoriasis treated for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic plaque psoriasis for at least 6 months
* Prior systemic therapy

Exclusion Criteria:

* Current or prior history of illness precluding use of immunomodulatory therapy.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 2004-12; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events
Abnormal laboratory values
Abnormal ECGs and vital signs

SECONDARY OUTCOMES:
PK/PD
Target lesion score after 28 days of treatment
Proportion of subjects meeting "clear" or "almost clear" criteria utilizing a static Physician's Global Assessment (sPGA)
Proportion of subjects demonstrating ≥ 50% and ≥ 75% decrease from baseline in Psoriasis Area and Severity Index (PASI) to the end of 28 days of treatment
Change in PASI from baseline to the end of 28 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kauffman, MD, PhD, Study Director — Vertex Pharmaceuticals Incorporated